CLINICAL TRIAL: NCT04085458
Title: Post-marketing Investigation (PMI) to Assess Safety and Efficacy of Jivi (BAY 94-9027) Treatment in Participants With Hemophilia A
Brief Title: Study to Gain More Information on How Safe and Effective Jivi Works in Patients With Severe Hemophilia A (Post-marketing Investigation)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19764; 2018-003655-37 (EudraCT Number)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Severe hemophilia A patients (Other): Prophylactic treatment regimens should be guided by clinical judgement based on individual patient characteristics and treatment response.
  Interventions: Drug: Damoctocog alfa pegol (Jivi, BAY94-9027)

INTERVENTIONS:
Drug: Damoctocog alfa pegol (Jivi, BAY94-9027) — The recommended starting dose is every 5 days treatment (45 IU/kg)- An assessment of response to treatment will be performed at the next scheduled visit after 10-15 ED (8-10 weeks). Participants may be assigned to different dosing regimens (every 7 days or 2x/week) or continue with every 5 days regimen, according to individual bleeding tendency and needs at investigator's discretion.

SUMMARY:
The goal of this study is to give gather more information on how safe and well Jivi works in patients with severe hemophilia A. Jivi has been approved by various regulatory agencies, including the FDA, Health Canada, Japanese Health Authority and the European Medicinal Agency. 25 patients will be enrolled and will stay for 1 to 2 years in this study depending on their treatment frequency. Researcher will monitor during the course of the study whether patients are developing antibodies (a protein made by the body in response to the drug) affecting the effectiveness of Jivi. In addition information on bleedings and patient's wellbeing will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participants must ≥ 18 years of age inclusive, at the time of signing the informed consent.
* Participants with severe hemophilia A (FVIII: C<1%)
* PTPs (Previously treated patients) (≥150 ED (Exposure day)) on prophylaxis treatment before enrollment
* Participants who are immunocompetent. If human immunodeficiency virus (HIV) positive, cluster of differentiation 4 (CD4)+ lymphocyte count >200/mm*3
* Participants who are willing to complete an eDiary
* Male participants
* Capable of giving signed informed consent

Exclusion Criteria:

* Any other inherited or acquired bleeding disorder in addition to Hemophilia A.
* Platelet count < 100,000/mm*3
* Creatinine > 2x upper limit of normal
* AST or ALT > 5x upper limit of normal (AST: aspartate aminotransferase; ALT: alanine aminotransferase)
* The participant has a planned major surgery.
* The participant is currently participating in another investigational drug study, or has participated in a clinical study involving an investigational drug within 30 days of signing informed consent or previous treatment in a clinical phase III study with BAY 94-9027 (now marketed as Jivi).
* Current evidence (by central laboratory) or history of inhibitor to FVIII with a titer ≥ 0.6 Bethesda unit (BU).
* Known hypersensitivity to the drug substance, excipients, or mouse or hamster protein.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Bulgaria (2):
  - UMHAT Tsaritsa Joanna-ISUL EAD Sofia, Sofia
  - MHAT Sveta Marina EAD, Varna
- Aarhus Universitetshospital, Skejby, Arhus N, Denmark
- LAIKO General Hospital of Athens, Athens, Greece
- Italy (3):
  - A.O. Pugliese-Ciaccio, Catanzaro, Calabria
  - A.O.U. Policlinico Umberto I, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
- Oslo Universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SP Szpital Kliniczny Nr 1, Wroclaw
- Spain (3):
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Universitario "La Paz", Madrid
  - Hospital Universitari i Politecnic La Fe | Hematologia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centers in 7 countries between 23 SEP 2019 (First participant first visit) and 26 Aug 2022 (last participant's data from the last visit were received). Bulgaria (2 centers), Denmark (1 centers), Spain (3 centers), Greece (1 center), Italy (3 centers), Norway (1 center), Poland (2 centers).
Pre-assignment Details: 36 participants were screened into the study (signed informed consent form (ICF)). 4 participants were screening failed.
Groups:
- Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment: Prophylaxis regimens with every 5 days treatment (45-60 IU/kg), or every 7 days (60 IU/kg) or twice per week (40 IU/kg).
Period: Overall Study
Arm/Group | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment
Started | 32
Completed | 27
Not Completed | 5
Not completed — Other | 1
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: FVIII Inhibitor Development by the Nijmegen Bethesda Assay
Description: FVIII inhibitor testing was performed using the Nijmegen-modified Bethesda assay. A positive inhibitor result was defined as a threshold of ≥0.6 BU/mL at the central laboratory and had to be confirmed with a second blood sample. After confirmation of the positive result, the inhibitor was to be reported as a serious adverse event (SAE).
Time Frame: Observed for 100 exposure days (EDs), up to 2 years
Population: Safety analysis set (SAF): A participant was included in the SAF if he received at least 1 infusion of study drug.
Measure: Number; unit: Participants
Arm/Group | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment
Number analyzed (Participants) | 32
Participants
  Any positive FVIII inhibitor | 0
  High titer FVIII inhibitor | 0
  Low titer FVIII inhibitor | 0

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-emergent AEs were defined as those that started after the first dose of study drug and up to 7 days after the last dose.
Time Frame: Observed for 100 exposure days (EDs), up to 2 years
Population: Safety analysis set (SAF): A participant was included in the SAF if he received at least 1 infusion of study drug.
Measure: Number; unit: participants
Arm/Group | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment
Number analyzed (Participants) | 32
participants
  Any AE | 21
  Any study drug-related AE | 3
  Any AE related to procedures required by the protocol | 0
  Any AE leading to discontinuation of study drug | 2
  Any SAE | 2
  Any study drug-related SAE | 0
  Any SAE related to procedures required by the protocol | 0
  Any SAE leading to discontinuation of study drug | 0
  AE with outcome death | 0

3. Secondary Outcome: Development of Treatment-emergent Anti-PEG Antibodies
Description: Anti-PEG antibody: antibody against the PEG moiety determined by enzyme-linked immunosorbent assay (ELISA). For participants with a positive result, IgM antibodies were tested.
Time Frame: Observed for 100 exposure days (EDs), up to 2 years
Population: Safety analysis set (SAF): A participant was included in the SAF if he received at least 1 infusion of study drug.
Measure: Number; unit: participants
Arm/Group | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment
Number analyzed (Participants) | 32
participants | 3

4. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: ABR is number of all bleeds per individual treatment period annualized to a 1-year time interval.
Time Frame: Observed for 100 exposure days (EDs), up to 2 years
Population: Modified intent-to-treat set (mITT): A participant was included in the mITT if he received at least 1 infusion of study drug and had injection/bleeding data available for at least 3 months. This time period is considered the minimum observation time for a reliable annualization of the observed bleed rate.
Measure: Median (Inter-Quartile Range); unit: Bleeds per year
Arm/Group | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment
Number analyzed (Participants) | 30
Bleeds per year | 1.8 [0.7 to 5.9]

ADVERSE EVENTS:
Time Frame: Timeframe for TEAEs: After the first study intervention up to 7 days after the end of study intervention, with an average of 475 days. Timeframe for the all-cause mortality: All deaths that occurred at any time during the study before the last contact, with an average of 476 days.
Arm/Group | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 15/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment (N=32)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Hemophilia A Patients With Damoctocog Alfa Pegol (Jivi, BAY94-9027) Treatment (N=32)
Pyrexia (General disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Tooth extraction (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT04085458/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT04085458/SAP_001.pdf